CLINICAL TRIAL: NCT03092726
Title: A Phase 2a, Randomized, Double-Blind Placebo-controlled, Parallel-group Study to Assess the Analgesic Efficacy and Safety of ASP8062 in Subjects With Fibromyalgia
Brief Title: A Study to Assess the Analgesic Efficacy and Safety of ASP8062 in Subjects With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8062-CL-0101
Record Dates: First submitted 2017-03-10; First posted 2017-03-28 (Actual); Results first posted 2019-03-28 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Fibromyalgia
Keywords: ASP8062; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — ASP8062

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP8062 (Experimental): Participants received 30 mg of ASP8062 orally once daily for 8 weeks.
  Interventions: Drug: ASP8062
- Placebo (Placebo Comparator): Participants received matching placebo orally once daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP8062 — ASP8062 30 mg was administered orally as a single daily dose, taken preferably in the morning with or without food.
  Arms: ASP8062
Drug: Placebo — Placebo was administered orally as a single daily dose, taken preferably in the morning with or without food.
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess analgesic efficacy of ASP8062 relative to placebo as well as the safety and tolerability. This study also assessed the treatment differences in physical function as well the improvements in overall subject status (e.g., fibromyalgia symptoms, global functioning) of ASP8062 relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) ≤ 45 kg/m^2.
* Female subject must either:

  * Be of nonchildbearing potential:
  * Postmenopausal (defined as at least 1 year without any menses) prior to Screening, or,
  * Documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy).
  * Or, if of childbearing potential, agree not to try to become pregnant during the study and for 28 days after the final study drug administration, have a negative blood pregnancy test at Screening and negative urine test on Day 1, and if heterosexually active, agree to consistently use 1 form of highly effective birth control starting at Screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must agree not to breastfeed at Screening and throughout the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at Screening, throughout the study period, and for 28 days after the final study drug administration.
* Male subject must not donate sperm starting at Screening and throughout the study period, and for 90 days after the final study drug administration.
* A sexually active male subject with female partner(s) who are of childbearing potential is eligible if:

  * Agree to use a male condom starting at screening and continue throughout study treatment and for 90 days after the final study drug administration. If the male subject has not had a vasectomy or is not sterile the male subjects female partner(s) is utilizing 1 form of highly effective birth control starting at screening and continue throughout study treatment, and for 90 days after the male subject receives final study drug administration.
* Male subject with a partner of child-bearing potential, or a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom throughout the study period and for 90 days after the final study drug administration.
* Subject meets the American College of Rheumatology (ACR) 1990 fibromyalgia diagnostic criteria at Screening:

  * Widespread pain for at least 3 months, defined as the presence of all of the following: Pain above and below the waist and pain in the axial skeleton (cervical spine or anterior chest or thoracic spine or low back) must be present.
  * Pain in at least 11 of 18 tender point sites on digital palpation. Digital palpation should be performed with an approximate force of 4 kg.
* Subject meets the ACR 2010 fibromyalgia diagnostic criteria at Screening:

  * Widespread pain index (WPI) ≥ 7 and symptom severity (SS) scale score ≥ 5 or WPI 3-6 and SS scale score ≥ 9.
  * Symptoms have been present at a similar level for at least 3 months.
  * The subject does not have a disorder that would otherwise explain the pain.
* Subject has a pain score ≥ 4 on the revised fibromyalgia impact questionnaire (FIQR) pain item at Screening.
* Subject is compliant with daily pain recordings during the Baseline Diary Run-In period, as defined by the completion of a minimum of 5 of 7 daily average pain ratings and agrees to complete daily diaries throughout the duration of the study.
* Subject has a mean daily average pain score ≥ 4 and ≤ 9 on an 11-point 0 to 10 NRS as recorded in the subject e-diary during the Baseline Diary Run-In period, and meeting pre-specified criteria for daily average pain scores.
* Subject agrees to use only acetaminophen as rescue medication for fibromyalgia pain throughout the course of the trial (up to 1000 mg per dose and not to exceed 3000 mg/day).
* Subject agrees not to initiate or change any non-pharmacologic interventions (including normal daily exercise routines, chiropractic care, physical therapy, psychotherapy, and massage therapy) during the course of the study. Non-pharmacologic interventions must be stable for a minimum of 30 days prior to Screening. And subject agrees to maintain usual level of activity for the duration of the study.
* Subject is capable of completing study assessments and procedures.
* Subject agrees not to participate in another interventional study from Screening through the End of Study (EOS) visit.

Exclusion Criteria:

* Subject has received an investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to Screening.
* Subject has had no meaningful improvement from 2 or more prior treatments (commercially available) for fibromyalgia (in at least 2 pharmacologic classes).
* Subject has had known hypersensitivity or intolerance to the use of acetaminophen or associated formulation components; known hypersensitivity to the formulation components of ASP8062.
* Subject has pain due to diabetic peripheral neuropathy, post-herpetic neuralgia, traumatic injury, prior surgery, complex regional pain syndrome, or other source of pain that would confound or interfere with the assessment of the subject's fibromyalgia pain or require excluded therapies during the subject's study participation.
* Subject has infectious or inflammatory arthritis (for example, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, gout), autoimmune disease (for example, systemic lupus erythematosus), or other widespread rheumatic disease other than fibromyalgia.
* Subject has a current, untreated moderate or severe major depressive disorder as assessed by the Mini-International Neuropsychiatric Interview (M.I.N.I.). Subject with current, treated major depressive disorder can be included provided that it is without clinically significant changes in symptoms while on the same dose of a protocol allowed antidepressant for greater than 60 days prior to Screening.
* Subject has initiated any non-pharmacologic interventions for the treatment of fibromyalgia or depression within 30 days prior to Screening or during the Screening period.
* Subject has a history of any psychotic and/or bipolar disorder as assessed by the M.I.N.I.
* Subject has a Hospital Anxiety and Depression Scale (HADS) score > 14 on the Depression subscale at Screening or at the time of Visit 3 (Randomization).
* Subject has a history of suicide attempt or suicidal behavior within the last 12 months, or has suicidal ideation within the last 12 months (a response of "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale C-SSRS]), or who is at significant risk to commit suicide at Screening and at the time of Visit 3 (Randomization).
* Subject has clinically significant abnormalities in clinical chemistry, hematology, or urinalysis, or a serum creatinine > 1.5 x the ULN at Screening. These assessments may be repeated once, after a reasonable time period (but within the Screening period).
* Subject has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 1.5 times the upper limit of the reference range at Screening. These assessments may be repeated once, after a reasonable time period (but within the Screening period).
* Subject has a positive test for hepatitis B surface antigen (HBsAg), hepatitis A virus antibodies (immunoglobulin M) (anti-HAV [IgM]) or hepatitis C virus antibodies (anti-HCV) at Screening or has history of a positive test for human immunodeficiency virus type 1(HIV-1) and/or type 2 (HIV-2).
* Subject has a resting systolic blood pressure > 180 mmHg or < 90 mmHg, and/or a sitting diastolic blood pressure > 100 mmHg at Screening. These assessments may be repeated once, after a reasonable time period (but within the Screening period).
* Subject has a clinically significant abnormality on 12-lead electrocardiogram (ECG) at Screening or Visit 3 (Randomization). If the ECG is abnormal an additional ECG can be carried out. If this also gives an abnormal result, the subject must be excluded.
* Subject has a history of myocardial infarction (within 6 months of Screening), unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsade de pointes, structural heart disease or a family history of Long QT Syndrome.
* Subject has evidence of any clinically significant, uncontrolled cardiovascular, gastrointestinal, endocrinologic (low thyroid stimulating hormone [TSH], but euthyroid is allowed), hematologic, hepatic, immunologic, infectious, metabolic, urologic, pulmonary (including obstructive sleep apnea not controlled by a continuous positive airway pressure device) neurologic, dermatologic, psychiatric, renal and/or other major disease (exclusive of fibromyalgia).
* Subject has planned surgery during the study participation.
* Subject has an active malignancy or a history of malignancy (except for treated nonmelanoma skin cancer) within 5 years of Screening.
* Subject has a positive drug or alcohol test at Screening, Baseline Diary Run-In or prior to Randomization. However, a positive test for tetrahydrocannabinol (THC) and/or opioids is allowed at the Screening visit, but must be confirmed negative prior to Baseline Diary Run-In and Randomization.
* Subject has a current or recent (within 12 months of Screening) history of a substance use disorder including cannabinoid and/or alcohol abuse disorder. Subject has used opioids for pain for more than 4 days during the week preceding the Screening visit.
* Subject is currently using protocol specified prohibited medications and is unable to wash-out including over-the-counter (OTC) products and grapefruit and/or grapefruit juice.
* Subject has filed or is awaiting judgment on a disability claim or has any pending worker's compensation litigation or related monetary settlements.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject is an employee of the Astellas Group, the Contract Research Organization (CRO) involved, or the investigator site personnel directly affiliated with this study and/or immediate families (spouse, parent, child, or sibling, whether biological or legally adopted).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (24):
- United States (24):
  - Noesis Pharma, LLC, Phoenix, Arizona
  - Excell Research, Inc, Oceanside, California
  - Collaborative Neuroscience Network, LLC., Torrance, California
  - PAB Clinical Research, Brandon, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Chicago Research Center, Inc, Chicago, Illinois
  - Medisphere Medical Research Center, LLC, Evansville, Indiana
  - Infinity Medical Research, Inc, North Dartmouth, Massachusetts
  - Elite Clinical Research, LLC, Jackson, Mississippi
  - The Center For Pharmaceutical Research, Kansas City, Missouri
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - NY Scientific, Brooklyn, New York
  - Neurobehavioral Research, Inc, Cedarhurst, New York
  - Private Practice, Raleigh, North Carolina
  - PMG of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Neuro-Behavioral Clinical Research, Inc, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Summit Research Network, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Clinical Investigation Specialists, Inc, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=338

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with fibromyalgia (FM) were enrolled in 24 sites in the United States.
Pre-assignment Details: Participants underwent a screening period (up to 42 days), where washout of medications and a 7-day baseline diary run-in were completed. Participants were randomized (1:1 ratio) after confirmation of eligibility (which also required a mean daily average pain score of ≥ 4 and ≤ 9 [per Daily Average Pain Numerical Rating Scale] to enter the study).
Period: Overall Study
Arm/Group | Placebo | ASP8062
Started | 88 | 95
Treated | 88 | 95
Completed (Completed the treatment period.) | 79 | 81
Not Completed | 9 | 14
Not completed — Adverse Event | 3 | 10
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Population: The analysis population was the safety analysis set (SAF), which consisted of all randomized participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ASP8062 | Total
Number analyzed (Participants) | 88 | 95 | 183
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 51.3 (12.9) | 52.5 (11.9) | 51.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 93 | 176
  Male | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 69 | 70 | 139
  Race: Black or African American | 15 | 20 | 35
  Race: Asian | 3 | 1 | 4
  Race: American Indian or Alaska Native | 0 | 3 | 3
  Race: Other | 1 | 1 | 2
Ethnicity [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 71 | 77 | 148
  Hispanic or Latino | 17 | 18 | 35
Baseline Mean Daily Average Pain Score Group [Count of Participants; unit: Participants] — The baseline mean daily average pain score was assessed through the Daily Average Pain NRS, which is a generic instrument for the assessment of pain that consists of a single question that asks participants to record their daily average pain on an 11-point scale, where 0 anchors "no pain" and 10 "pain as bad as you can imagine." The baseline mean daily average pain score was calculated from data recorded by participants in the 7-day electronic baseline diary. Population: The analysis population was the FAS.
  Participants
    No pain: 0 | 0 | 0 | 0
    Mild: > 0 to < 4 | 0 | 0 | 0
    Moderate: >= 4 to < 7 | 59 | 57 | 116
    Severe: >= 7 to 10 | 29 | 38 | 67
Baseline Mean Daily Average Pain Score [Mean (Standard Deviation); unit: units on a scale] — The baseline mean daily average pain score was assessed through the Daily Average Pain NRS, which is a generic instrument for the assessment of pain that consists of a single question that asks participants to record their daily average pain on an 11-point scale, where 0 anchors "no pain" and 10 "pain as bad as you can imagine." The baseline mean daily average pain score was calculated from data recorded by participants in the 7-day electronic baseline diary. Population: The analysis population was the full analysis set (FAS), which consisted of all randomized participants who took at least 1 dose of study drug.
  units on a scale | 6.49 (1.03) | 6.54 (0.97) | 6.51 (1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Mean Daily Average Pain Score as Assessed by Numerical Rating Scale (NRS)
Description: The mean daily average pain score was assessed thorugh the Daily Average Pain NRS, which is a generic instrument for the assessment of pain that consists of a single question that asks participants to record their daily average pain on an 11-point scale, where 0 anchors "no pain" and 10 "pain as bad as you can imagine." The mean daily average pain score was calculated from data recorded by participants daily in the electronic diary, and the recall period was the last 24 hours. A negative change indicated a reduction/improvement from baseline (i.e., a favorable outcome).
Time Frame: Baseline and week 8
Population: The analysis population was the full analysis set (FAS), which consisted of all randomized participants who took at least 1 dose of study drug. Participants with available data at baseline were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | ASP8062
Number analyzed (Participants) | 88 | 95
Units on a scale | -1.42 (0.19) | -1.36 (0.19)
Statistical Analysis 1: Comparison: Placebo vs ASP8062; Differences of least squares (LS) means were calculated by subtracting the LS mean of placebo group from the LS mean of ASP8062 30 mg group using a mixed-effect, repeated measures (MMRM) model with change from baseline to each week from weeks 1 to 8 as response, treatment, center (pooled where necessary), time (study weeks 1 to 8) and treatment-by-time interaction as fixed effects, baseline and baseline-by-time interaction as covariates; Test type: Superiority; p = 0.590, MMRM — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described MMRM model; LS Mean (LSM) Difference = 0.06, 90% CI 2-sided [-0.38 to 0.50], Standard Error of Mean 0.26

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Safety was assessed by adverse events (AEs), which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study drug or was clinically significant. A TEAE was defined as any AE that started or worsened after the first dose of study drug up to 30 days after the last dose of study drug. AEs were considered serious (SAEs) if the AE resulted in death, was life-threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly, or birth defect or required inpatient hospitalization or led to prolongation of hospitalization. TEAEs in drug abuse, dependence and withdrawal standardized MedDRA query (SMQ) are special AEs of interest grouped together using the SMQ tool (MedDRA v20.0).
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to 87 days)
Population: The analysis population was the SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ASP8062
Number analyzed (Participants) | 88 | 95
Participants
  Any TEAE | 43 | 67
  Drug-related TEAE | 19 | 45
  Serious TEAE | 0 | 0
  Drug-related serious TEAE | 0 | 0
  TEAE leading to withdrawal of treatment | 3 | 10
  Death | 0 | 0
  TEAE in drug abuse, dependence, withdrawal SMQ | 0 | 0
  TEAE in drug abuse and dependence SMQ | 0 | 0
  TEAE in drug withdrawal SMQ | 0 | 0
  Drug abuse-related TEAEs | 0 | 1
  Drug withdrawal-related TEAEs | 18 | 26

3. Primary Outcome: Number of Participants With an Affirmative Response to Columbia Suicide Severity Rating Scale (C-SSRS): Suicidal Ideation
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) is a questionnaire used for suicide risk assessment. Affirmative or negative responses were provided to 5 items to suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent).
Time Frame: Weeks 1 to 8
Population: The analysis population was the SAF. Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ASP8062
Number analyzed (Participants) | 86 | 90
Participants
  Wish to be dead | 1 | 1
  Non-specific active suicidal thoughts | 0 | 0
  With any methods (not plan) w/o intent to act | 0 | 0
  With some intent to act, w/o specific plan | 0 | 0
  With specific plan and intent | 0 | 0

4. Primary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Behavior
Description: The C-SSRS is a questionnaire used for suicide risk assessment. Affirmative or negative responses were provided to 5 items to suicidal behavior (1. Preparatory acts or behavior, 2. Aborted attempt, 3. Interrupted attempt, 4. Actual attempt, 5. Completed suicide).
Time Frame: Weeks 1 to 8
Population: The analysis population was the SAF. Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ASP8062
Number analyzed (Participants) | 86 | 90
Participants
  Preparatory acts or behavior | 0 | 0
  Aborted attempt | 0 | 0
  Interrupted attempt | 0 | 0
  Actual attempt | 0 | 0
  Completed suicide | 0 | 0

5. Secondary Outcome: Percentage of Participants With ≥ 30% Reduction From Baseline to Week 8 and End of Treatment (EOT) in Mean Daily Average Pain Score as Assessed by NRS
Description: The mean daily average pain score was assessed through the Daily Average Pain NRS, which is a generic instrument for the assessment of pain that consists of a single question that asks participants to record their daily average pain on an 11-point scale, where 0 anchors "no pain" and 10 "pain as bad as you can imagine." The mean daily average pain score was calculated from data recorded by participants daily in the electronic diary, and the recall period was the last 24 hours. For the week 8 analysis, participants with missing baseline or week 8 data were classified as nonresponders. For EOT analysis, participants with missing baseline or EOT data were classified as nonresponders.
Time Frame: Baseline to week 8
Population: The analysis population was the FAS. Baseline Observation Carried Forward (BOCF) was used for week 8. Last Observation Carried Forward (LOCF) was used for EOT.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ASP8062
Number analyzed (Participants) | 88 | 95
Percentage of participants
  Week 8 | 31.8 [23.6 to 40.9] | 25.3 [18.1 to 33.7]
  EOT | 33.0 [24.7 to 42.1] | 27.4 [19.9 to 35.9]
Statistical Analysis 1: Comparison: Placebo vs ASP8062; Week 8: Differences of the percentages were calculated by subtracting the percentage of placebo group from the percentage of ASP8062 30 mg group. Confidence Interval (CI) for each treatment group and the difference of the percentages was an exact unconditional confidence interval based on Santner-Snell approach; Test type: Superiority; p = 0.874, Fisher Exact — 1-sided p-value is for comparison of ASP8062 30 mg with placebo using Fisher's Exact method; Difference of percentages = -6.6, 90% CI 2-sided [-18.7 to 5.7]
Statistical Analysis 2: Comparison: Placebo vs ASP8062; EOT: Differences of the percentages were calculated by subtracting the percentage of placebo group from the percentage of ASP8062 30 mg group. Confidence Interval (CI) for each treatment group and the difference of the percentages was an exact unconditional confidence interval based on Santner-Snell approach; Test type: Superiority; p = 0.838, Fisher Exact — 1-sided p-value is for comparison of ASP8062 30 mg with placebo using Fisher's Exact method; Differences of percentages = -5.6, 90% CI 2-sided [-17.7 to 6.7]

6. Secondary Outcome: Percentage of Participants With ≥ 50% Reduction From Baseline to Week 8 and EOT in Mean Daily Average Pain Score as Assessed by NRS
Description: The mean daily average pain score was assessed thorugh the Daily Average Pain NRS, which is a generic instrument for the assessment of pain that consists of a single question that asks participants to record their daily average pain on an 11-point scale, where 0 anchors "no pain" and 10 "pain as bad as you can imagine." The mean daily average pain score was calculated from data recorded by participants daily in the electronic diary, and the recall period was the last 24 hours. For the week 8 analysis, participants with missing baseline or week 8 data were classified as nonresponders. For EOT analysis, participants with missing baseline or EOT data were classified as nonresponders.
Time Frame: Baseline to week 8
Population: The analysis population was the FAS. BOCF was used for week 8. LOCF was used for EOT.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ASP8062
Number analyzed (Participants) | 88 | 95
Percentage of participants
  Week 8 | 12.5 [7.2 to 19.8] | 14.7 [9.1 to 22.1]
  EOT | 12.5 [7.2 to 19.8] | 16.8 [10.9 to 24.4]
Statistical Analysis 1: Comparison: Placebo vs ASP8062; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.412, Fisher Exact — 1-sided p-value is for comparison of ASP8062 30 mg with placebo using Fisher's Exact method; Differences of percentages = 2.2, 90% CI 2-sided [-10.0 to 14.4]
Statistical Analysis 2: Comparison: Placebo vs ASP8062; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.269, Fisher Exact — 1-sided p-value is for comparison of ASP8062 30 mg with placebo using Fisher's Exact method; Differences of percentages = 4.3, 90% CI 2-sided [-7.9 to 16.4]

7. Secondary Outcome: Change From Baseline to Weeks 2, 4, 8 and EOT in the Fibromyalgia Impact Questionnaire Revised (FIQR) Function Subscale Score
Description: The FIQR was developed to capture total spectrum of problems related to fibromyalgia and the responses to therapy. The 21-item FIQR contains 3 subscales: function (9 questions), overall impact (2 questions), and symptoms (10 questions). Participants answer each question on an 11-point NRS, with anchors appropriate to each question on a tablet device during a visit. The recall period was the last 7 days or the last time the activity was performed if not within the 7-day recall period. The Function subscale has a range of scores of 0 to 90, with a lower score indicating better (higher) function. A negative change indicated a reduction/improvement from baseline (i.e., a favorable outcome).
Time Frame: Baseline and weeks 2, 4, 8
Population: The analysis population was the FAS. Participants with available data at baseline were included in the analysis. LOCF was used for EOT.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | ASP8062
Number analyzed (Participants) | 88 | 95
Units on a scale
  Week 2: number analyzed (Participants) | 86 | 90
  Week 2 | -8.21 (1.46) | -8.89 (1.42)
  Week 4: number analyzed (Participants) | 83 | 82
  Week 4 | -10.25 (1.67) | -10.89 (1.65)
  Week 8: number analyzed (Participants) | 80 | 79
  Week 8 | -12.88 (1.91) | -12.02 (1.89)
  EOT | -12.05 (1.87) | -10.96 (1.78)
Statistical Analysis 1: Comparison: Placebo vs ASP8062; Week 2: Differences of LS means were calculated by subtracting the LS mean of placebo group from the LS mean of ASP8062 30 mg group using a MMRM model with change from baseline to weeks 2, 4 and 8 as response, treatment, center (pooled where necessary), time (study weeks 2, 4 and 8) and treatment-by-time interaction as fixed effects, baseline and baseline-by-time interaction as covariates; Test type: Superiority; p = 0.369, MMRM — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described MMRM model; LSM Difference = -0.68, 90% CI 2-sided [-4.05 to 2.68], Standard Error of Mean 2.03
Statistical Analysis 2: Comparison: Placebo vs ASP8062; Week 4: Differences of LS means were calculated by subtracting the LS mean of placebo group from the LS mean of ASP8062 30 mg group using a MMRM model with change from baseline to weeks 2, 4 and 8 as response, treatment, center (pooled where necessary), time (study weeks 2, 4 and 8) and treatment-by-time interaction as fixed effects, baseline and baseline-by-time interaction as covariates; Test type: Superiority; p = 0.393, MMRM — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described MMRM model; LSM Difference = -0.64, 90% CI 2-sided [-4.51 to 3.24], Standard Error of Mean 2.34
Statistical Analysis 3: Comparison: Placebo vs ASP8062; Week 8: Differences of LS means were calculated by subtracting the LS mean of placebo group from the LS mean of ASP8062 30 mg group using a MMRM model with change from baseline to weeks 2, 4 and 8 as response, treatment, center (pooled where necessary), time (study weeks 2, 4 and 8) and treatment-by-time interaction as fixed effects, baseline and baseline-by-time interaction as covariates; Test type: Superiority; p = 0.626, MMRM; LSM Difference = 0.86, 90% CI 2-sided [-3.57 to 5.30], Standard Error of Mean 2.68
Statistical Analysis 4: Comparison: Placebo vs ASP8062; EOT: Differences of LS means were calculated by subtracting the LS mean of placebo group from the LS mean of ASP8062 30 mg group using an ANCOVA model that was performed with change from baseline at the EOT timepoint as response, treatment and center (pooled where necessary) as fixed effects and baseline as a covariate; Test type: Superiority; p = 0.664, ANCOVA — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described ANCOVA model; LSM Difference = 1.09, 90% CI 2-sided [-3.16 to 5.34], Standard Error of Mean 2.57

8. Secondary Outcome: Change From Baseline to Weeks 2, 4, 8, and EOT in the FIQR Symptoms Subscale Score
Description: The FIQR was developed to capture the total spectrum of problems related to fibromyalgia and the responses to therapy. The 21-item FIQR contains 3 subscales: function (9 questions), overall impact (2 questions), and symptoms (10 questions). Participants answer each question on an 11-point NRS, with anchors appropriate to each question on a tablet device during a visit. The recall period was the last 7 days. The Symptoms subscale range of scores is 0 to 100, with a lower score indicating a better (lower) level of symptoms. A negative change indicates a reduction/improvement from baseline (i.e., a favorable outcome).
Time Frame: Baseline and weeks 2, 4, 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | ASP8062
Number analyzed (Participants) | 88 | 95
Units on a scale
  Week 2: number analyzed (Participants) | 86 | 90
  Week 2 | -9.05 (1.33) | -8.89 (1.29)
  Week 4: number analyzed (Participants) | 83 | 82
  Week 4 | -10.91 (1.49) | -9.45 (1.46)
  Week 8: number analyzed (Participants) | 80 | 79
  Week 8 | -12.40 (1.83) | -10.70 (1.82)
  EOT | -11.47 (1.77) | -9.79 (1.69)
Statistical Analysis 1: Comparison: Placebo vs ASP8062; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.534, MMRM — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described MMRM model; LSM Difference = 0.16, 90% CI 2-sided [-2.90 to 3.22], Standard Error of Mean 1.85
Statistical Analysis 2: Comparison: Placebo vs ASP8062; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.758, MMRM — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described MMRM model; LSM Difference = 1.46, 90% CI 2-sided [-1.98 to 4.91], Standard Error of Mean 2.08
Statistical Analysis 3: Comparison: Placebo vs ASP8062; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.745, MMRM — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described MMRM model; LSM Difference = 1.70, 90% CI 2-sided [-2.56 to 5.96], Standard Error of Mean 2.57
Statistical Analysis 4: Comparison: Placebo vs ASP8062; [analysis description as in outcome 7, analysis 4]; Test type: Superiority; p = 0.755, ANCOVA — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described ANCOVA model; LSM Difference = 1.68, 90% CI 2-sided [-2.34 to 5.69], Standard Error of Mean 2.43

9. Secondary Outcome: Change From Baseline to Weeks 2, 4, 8, and EOT in the FIQR Overall Impact Subscale Score
Description: The FIQR was developed to capture the total spectrum of problems related to fibromyalgia and the responses to therapy. The 21-item FIQR contains 3 subscales: function (9 questions), overall impact (2 questions), and symptoms (10 questions). Participants answer each question on an 11-point NRS, with anchors appropriate to each question on a tablet device during a visit. The recall period was the last 7 days. The Overall Impact subscale has a range of scores from 0 to 20, with a lower score indicating better (lower) impact. A negative change indicated a reduction/improvement from baseline (i.e., a favorable outcome).
Time Frame: Baseline and weeks 2, 4, 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | ASP8062
Number analyzed (Participants) | 88 | 95
Units on a scale
  Week 2: number analyzed (Participants) | 86 | 90
  Week 2 | -2.79 (0.42) | -2.60 (0.41)
  Week 4: number analyzed (Participants) | 83 | 82
  Week 4 | -3.04 (0.52) | -3.20 (0.51)
  Week 8: number analyzed (Participants) | 80 | 79
  Week 8 | -3.50 (0.50) | -3.44 (0.50)
  EOT | -3.38 (0.49) | -3.21 (0.46)
Statistical Analysis 1: Comparison: Placebo vs ASP8062; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.629, MMRM — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described MMRM model; LSM Difference = 0.19, 90% CI 2-sided [-0.78 to 1.17], Standard Error of Mean 0.59
Statistical Analysis 2: Comparison: Placebo vs ASP8062; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.410, MMRM — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described MMRM model; LSM Difference = -0.17, 90% CI 2-sided [-1.37 to 1.04], Standard Error of Mean 0.73
Statistical Analysis 3: Comparison: Placebo vs ASP8062; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.531, MMRM — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described MMRM model; LSM Difference = 0.06, 90% CI 2-sided [-1.11 to 1.22], Standard Error of Mean 0.71
Statistical Analysis 4: Comparison: Placebo vs ASP8062; [analysis description as in outcome 7, analysis 4]; Test type: Superiority; p = 0.603, ANCOVA — 1-sided p-value is for comparison of ASP8062 30 mg with placebo from the above described ANCOVA model; LSM Difference = 0.17, 90% CI 2-sided [-0.93 to 1.28], Standard Error of Mean 0.67

10. Secondary Outcome: Overall Participant Improvement as Assessed by Patient Global Impression of Change (PGIC)
Description: The PGIC is a self-administered 7-point Likert scale that asks participants to evaluate their fibromyalgia relative to baseline. This is a single question and the grade ranges from 1 ("Very Much Improved") to 7 ("Very Much Worse").
Time Frame: Weeks 2, 4, 8
Population: The analysis population was the FAS. Modified LOCF (mLOCF) was used for weeks 2, 4, and 8, where "No Change" was imputed for participants who discontinued due to lack of efficacy or AEs, and LOCF was used for participants who discontinued due to other reasons. LOCF was used for EOT.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ASP8062
Number analyzed (Participants) | 88 | 95
Participants
  Week 2: Very Much Improved | 0 | 4
  Week 2: Much Improved | 7 | 9
  Week 2: Minimally Improved | 34 | 28
  Week 2: No Change | 34 | 42
  Week 2: Minimally Worse | 7 | 9
  Week 2: Much Worse | 5 | 3
  Week 2: Very Much Worse | 1 | 0
  Week 4: Very Much Improved | 2 | 6
  Week 4: Much Improved | 13 | 13
  Week 4: Minimally Improved | 34 | 23
  Week 4: No Change | 28 | 39
  Week 4: Minimally Worse | 8 | 6
  Week 4: Much Worse | 3 | 8
  Week 4: Very Much Worse | 0 | 0
  Week 8: Very Much Improved | 5 | 12
  Week 8: Much Improved | 13 | 12
  Week 8: Minimally Improved | 33 | 17
  Week 8: No Change | 26 | 38
  Week 8: Minimally Worse | 6 | 10
  Week 8: Much Worse | 4 | 6
  Week 8: Very Much Worse | 1 | 0
  EOT: Very Much Improved | 5 | 12
  EOT: Much Improved | 13 | 12
  EOT: Minimally Improved | 34 | 19
  EOT: No Change | 24 | 34
  EOT: Minimally Worse | 6 | 11
  EOT: Much Worse | 4 | 7
  EOT: Very Much Worse | 2 | 0
Statistical Analysis 1: Comparison: Placebo vs ASP8062; Week 2: Odds ratio of ASP8062 30 mg versus placebo, associated 90% 2-sided CI and p-value was estimated using a proportional odds model including treatment group as a factor; Test type: Superiority; p = 0.811, Proportional Odds model — 2-sided p-value is for the comparison of ASP8062 30 mg with placebo from the above described proportional odds model; Odds Ratio (OR) = 1.07, 90% CI 2-sided [0.68 to 1.67]
Statistical Analysis 2: Comparison: Placebo vs ASP8062; Week 4: Odds ratio of ASP8062 30 mg versus placebo, associated 90% 2-sided CI and p-value was estimated using a proportional odds model including treatment group as a factor; Test type: Superiority; p = 0.368, Proportional Odds model — 2-sided p-value is for the comparison of ASP8062 30 mg with placebo from the above described proportional odds model; Odds Ratio (OR) = 0.79, 90% CI 2-sided [0.50 to 1.22]
Statistical Analysis 3: Comparison: Placebo vs ASP8062; Week 8: Odds ratio of ASP8062 30 mg versus placebo, associated 90% 2-sided CI and p-value was estimated using a proportional odds model including treatment group as a factor; Test type: Superiority; p = 0.357, Proportional Odds model — 2-sided p-value is for the comparison of ASP8062 30 mg with placebo from the above described proportional odds model; Odds Ratio (OR) = 0.78, 90% CI 2-sided [0.50 to 1.21]
Statistical Analysis 4: Comparison: Placebo vs ASP8062; EOT: Odds ratio of ASP8062 30 mg versus placebo, associated 90% 2-sided CI and p-value was estimated using a proportional odds model including treatment group as a factor; Test type: Superiority; p = 0.407, Proportional Odds model — 2-sided p-value is for the comparison of ASP8062 30 mg with placebo from the above described proportional odds model; Odds Ratio (OR) = 0.80, 90% CI 2-sided [0.52 to 1.24]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to 87 days)
Groups:
- ASP8062 30 mg: Participants received 30 mg of ASP8062 orally once daily for 8 weeks.
Arm/Group | Placebo | ASP8062 30 mg
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/95
Other Adverse Events (participants affected / at risk) | 17/88 | 38/95
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=88) | ASP8062 30 mg (N=95)
Nausea (Gastrointestinal disorders) | 4 (5) | 6 (6)
Urinary tract infection (Infections and infestations) | 5 (5) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 28 (33)
Headache (Nervous system disorders) | 10 (11) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03092726/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT03092726/SAP_001.pdf